CLINICAL TRIAL: NCT06949293
Title: The Effect of Classical Hand Massage, Lavender Inhalation and Hand Massage With Lavender on Anxiety, Pain and Comfort in Patients Undergoing Cystoscopy
Brief Title: The Effect of Classical Hand Massage, Lavender Inhalation and Hand Massage With Lavender on Anxiety, Pain and Comfort
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afide Tufan (Other)
Responsible Party: Sponsor-Investigator, Afide Tufan, Principal Investigator, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-10840098-202.3.02-3033
Record Dates: First submitted 2025-04-12; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cystoscopy; Aromatherapy; Hand Massage
Keywords: Aromatherapy; Pain; Anxiety; Hand Massage; Comfort; Cystoscopy
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — lavender oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Classic hand massage group (Active Comparator): Patients included in the study who are planned to undergo cystoscopy will be assigned to the classical hand massage group by matching them with the randomization table according to the order of arrival. There will be 36 patients in this group.
  Interventions: Other: Classic hand massage
- Lavender inhalation group (Active Comparator): Patients included in the study who are planned to undergo cystoscopy will be assigned to the lavender inhalation group by matching them with the randomization table according to the order of arrival. There will be 36 patients in this group.
  Interventions: Other: Lavender inhalation
- Hand massage group with lavender oil (Active Comparator): The patients included in the study who are planned to undergo cystoscopy will be assigned to the hand massage group with lavender oil by matching them with the randomization table according to the order of arrival. There will be 36 patients in this group.
  Interventions: Other: Hand massage with lavender oil
- Control group (No Intervention): This group will not receive any intervention other than routine practice. There will be 36 patients in this group.

INTERVENTIONS:
Other: Hand massage with lavender oil — Each hand of the patient will be massaged with lavender oil for 5 minutes before and during cystoscopy. Before the application, 5% lavender oil will be applied to a small part of the hand and this area will be monitored for signs of allergic reaction such as swelling and redness. If no allergic reaction is observed, the study will continue.
  Arms: Hand massage group with lavender oil
Other: Classic hand massage — Each hand of the patient will be massaged with baby oil for 5 minutes before and during the cystoscopy procedure.
  Arms: Classic hand massage group
Other: Lavender inhalation — Before and during the cystoscopy procedure, 2-3 drops of 5% lavender oil will be poured onto a 5x5 cm sterile gauze. It will be placed 10 cm away from the patient's nose and sniffed for 10 minutes.
  Arms: Lavender inhalation group

SUMMARY:
Cystoscopy is one of the most commonly performed urologic procedures to examine the anatomy and evaluate pathologies of the lower urinary tract. Although cystoscopy is a safe procedure with a low risk of morbidity, it can often cause pain, anxiety and restlessness in patients. This study aims to determine the effects of classical hand massage, lavender inhalation and lavender hand massage applied to patients undergoing cystoscopy on the patient's anxiety, pain and comfort. The population of the study will consist of patients who underwent cystoscopy between July 2024 and April 2025. Data will be obtained with the Patient Identification Form, Vital Signs Follow-up Form, State Anxiety Scale, Numerical Pain Scale and Numerical Comfort Scale. The research will be conducted in three stages: before, during and after the cystoscopy procedure. In the pre-cystoscopy period, patients who meet the study inclusion criteria will be informed about the procedure and verbal and written permissions will be obtained. Randomization will be performed according to the order of application and the patients will be divided into four groups as the classical hand massage group, the lavender inhalation group, the lavender hand massage group and the control group. The Patient Identification Form will be filled in and the scales will be introduced. The vital signs of the patients in the intervention groups will be assessed half an hour before the procedure and the State Anxiety Scale will be filled in. In addition, a ten-minute application will be performed before the procedure and their vital signs and the State Anxiety Scale will be assessed five minutes after the procedure. During the cystoscopy period, after the patients in the intervention group are taken to the cystoscopy table and lidocaine gel is applied, their vital signs and pain levels will be assessed during the passage of the cystoscopy instrument from the urethra to the bladder. A ten-minute application will be performed during the procedure in the intervention groups and their vital signs and pain will be assessed immediately after the cystoscopy is completed. In the post-procedure period, half an hour after the cystoscopy procedure, the vital signs of the patients will be measured again, and the Numerical Pain Scale and Numerical Comfort Scale will be filled. The same data will be collected from the patients in the control group without any application.

DETAILED DESCRIPTION:
Cystoscopy is one of the most commonly performed urological procedures to evaluate lower urinary tract symptoms such as hematuria and urinary incontinence as well as various pathologies of the urethra, prostate and bladder and to examine the anatomy of the lower urinary tract. Although cystoscopy is a safe procedure with a low risk of morbidity, it is invasive and can be associated with pain and anxiety. Cystoscopy is performed after a standard physical examination, disinfection of the external genital organs and instillation of some kind of lubricant into the urethra. In the majority of cases, general anesthesia is not required and it is performed under sedation or local anesthesia.However, some studies have shown that many patients report that they still feel pain during the procedure, although not at an uncomfortable level and for different reasons. Male patients are reported to experience more pain with rigid cystoscopy, first-time cystoscopies and cystoscopies to investigate lower urinary tract symptoms. Although cystoscopy is generally well tolerated, some patients describe the pain associated with the procedure as "excruciating".

Cystoscopy can often cause anxiety and discomfort. Especially in conscious patients, direct exposure to various stimuli during cystoscopy increases anxiety. Pain and anxiety associated with cystoscopy can activate the sympathetic nervous system, resulting in a variety of physiologic responses, including increased cardiac output, elevated blood glucose levels, peripheral vascular contraction, and elevated blood pressure.Often acute pain causes anxiety, which increases fear of pain and depression, sleep disturbances, and interferes with concentration and cognition. Anxiety about pain causes individuals to avoid the stimulus and overreact to the accompanying body sensations. Ensuring the comfort of patients before, during and after the cystoscopy procedure is necessary and important for the quality of care. Patients may experience discomfort and restlessness due to anxiety and stress. More than half of patients undergoing cystoscopy report moderate to severe discomfort, which is a significant problem for patients undergoing the procedure. It has also been found that men experience more discomfort than women.

There are various strategies to reduce anxiety and pain, including pharmacologic and nonpharmacologic methods. Although lidocaine lubricants, pain medications or flexible cystoscopy can be used to alleviate pain and anxiety during cystoscopy, the procedure still causes discomfort. Therefore, non-pharmacologic methods are needed to reduce pain and anxiety during the procedure and increase patient comfort and satisfaction. Non-pharmacological methods include aromatherapy, massage therapy, music therapy, hand holding, etc., which can be used alone or in combination with other methods. The advantages of these non-pharmacologic methods are that they are inexpensive, non-invasive, easy to apply and do not have chemical side effects.When the studies evaluating nursing care for the negative situations experienced by patients during cystoscopy were examined, it was found that listening to music during the procedure reduced patients' feelings of anxiety, pain, discomfort and dissatisfaction. There are also studies showing that the use of a virtual reality application during cystoscopy shortens the procedure time and reduces pain and discomfort. Hand holding during cystoscopy has also been shown to reduce patients' anxiety, pain and dissatisfaction. A study showed that watching relaxing videos during the procedure decreased pain, anxiety and hemodynamic parameters of female patients and increased their satisfaction levels. In another study conducted on women undergoing cystoscopy, it was determined that when patients' emotional, physical and informational needs were met, when they actively participated in their health care, when they had a say in their care, their fear of the unknown decreased and patient satisfaction increased.

In this study, the effect of classical hand massage, lavender inhalation and hand massage with lavender on reducing the anxiety of the patients before the cystoscopy procedure and the effect of the interventions during the procedure on reducing pain and increasing comfort will be evaluated. When the literature was examined, it was found that non-pharmacologic interventions applied during cystoscopy included distraction methods such as listening to music, virtual reality, watching relaxing videos, and squeezing a stress ball. There is no study showing whether classical hand massage, lavender inhalation and hand massage with lavender are effective in affecting the patient's anxiety, pain and comfort in patients undergoing cystoscopy. This study will be a first in this context. If the interventions applied to the intervention group are found to be effective, they can be recommended as methods that can be used routinely before and during the cystoscopy procedure. With this study, it is aimed to reduce the level of anxiety before cystoscopy procedure, to reduce pain during and after the procedure and to contribute to increase comfort.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Being a man
* Having cystoscopy for the first time,
* Local anesthesia will be performed,
* Rigid cystoscopy will be performed,
* No obstacles to communication,
* Having a good sense of smell,
* No known history of allergy to the essential oil used,
* To agree to participate in the research

Exclusion Criteria:

* Having any contraindication for the procedure (urinary tract infection, lidocaine allergy, anatomical problems with the urethra, etc.),
* Having used any painkiller at least 24 hours before cystoscopy,
* Performing manipulations such as bladder biopsy, Double J catheter insertion or removal

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
participants' level of anxiety | Perioperative
  State Anxiety Scale:The scale developed by Spielberg et al. in 1964 to measure the state anxiety levels of normal and abnormal individuals was adapted into Turkish by Öner and Le Compte (1983). It is a self-assessment type scale consisting of short statements. It was developed to measure a person's anxiety at a particular moment. The state anxiety scale, which consists of 20 items, is a scale that determines how an individual feels at a particular moment and condition. The emotions or behaviors expressed in the items of the SCS are answered by marking one of the options according to the degree of intensity (1) not at all, (2) a little, (3) a lot, (4) completely. There are 10 reversed statements in the inventory. These statements are items 1,2,5,8,10,11,15,16,19 and 20. The state anxiety score is calculated by adding 50 points to the difference between the total weighted scores of the direct and inverted statements. The scores obtained in the state anxiety scale theoretically vary betw
participants' level of pain | Perioperative
  Numeric Pain Scale: This scale, which is intended to determine the severity of pain, aims to explain the patient's pain with numbers. The "0-10" numerical pain scale was used to assess the severity of the patients' pain. On numerical scales, pain starts with absence of pain (0) and reaches up to unbearable pain (10).
Number of Participants with high comfort rate | Perioperative
  Numerical Comfort Scale: It is a 10 cm long, horizontally usable measurement tool for determining the comfort level, starting with "0- most uncomfortable" and ending with "10- most comfortable". A high score indicates a high comfort level
Body temperature of participants | Perioperative
  The researcher will be measured with a digital non-contact thermometer.
Systolic and diastollic blood pressure of participants | Perioperative
  The researcher will measure it using a digital blood pressure monitor.
Pulse rate of participants | Perioperative
  The researcher will measure it using pulse oximetry
Oxygen saturation of participants | Perioperative
  The researcher will measure it using pulse oximetry

CONTACTS AND LOCATIONS:
Overall Officials: Selda RIZALAR, Prof. Dr., Study Director — The University of Health Sciences
Locations (1):
- Kula State Hospital, Manisa, Kula, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwon WA, Lee JW, Seo HK, Oh TH, Park SC, Jeong HJ, Seo IY. Hand-Holding during Cystoscopy Decreases Patient Anxiety, Pain, and Dissatisfaction: A Pilot Randomized Controlled Trial. Urol Int. 2018;100(2):222-227. doi: 10.1159/000485745. Epub 2017 Dec 22. PMID 29275402
- [Background] Krajewski W, Zdrojowy R, Wojciechowska J, Koscielska K, Dembowski J, Matuszewski M, Tupikowski K, Malkiewicz B, Kolodziej A. Patient comfort during flexible and rigid cystourethroscopy. Wideochir Inne Tech Maloinwazyjne. 2016;11(2):94-7. doi: 10.5114/wiitm.2016.60665. Epub 2016 Jun 17. PMID 27458489
- [Background] Laszkiewicz J, Krajewski W, Luczak M, Chorbinska J, Nowak L, Bardowska K, Zdrojowy R. Pain reduction methods during transurethral cystoscopy. Contemp Oncol (Pozn). 2021;25(2):80-87. doi: 10.5114/wo.2021.106652. Epub 2021 May 28. PMID 34667433
- [Background] Gezginci E, Bedir S, Ozcan C, Iyigun E. Does Watching a Relaxing Video During Cystoscopy Affect Pain and Anxiety Levels of Female Patients? A Randomized Controlled Trial. Pain Manag Nurs. 2021 Apr;22(2):214-219. doi: 10.1016/j.pmn.2020.08.005. Epub 2020 Sep 29. PMID 33008780